CLINICAL TRIAL: NCT01907919
Title: Diode Laser-Assisted Direct Pulp Capping In Permanent Teeth
Brief Title: Pilot Study,Diode Laser 808 nm Supported Direct Pulp Capping in Permanent Teeth
Acronym: Laser in DPC
Status: Completed | Type: Observational
Sponsor: Yazdanfar, Iraj, M.D. (Individual)
Collaborators: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, iraj yazdanfar, M.Sc in laser in dentistry, Yazdanfar, Iraj, M.D.
Other Study IDs: private practice
Record Dates: First submitted 2013-07-12; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Haemostatic; Bacterial De-contamination; Bio-stimulation; Reparative Dentine Formation; Pain Reduction
Keywords: Pulp capping, Diode laser 808 nm, Tertiary dentin, RM-GIC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

GROUPS / COHORTS (2):
- conventional group,RM-GIC: 1. Group A: Five teeth were treated with traditional rotating instruments, the cavities were prepared with diamond drills by turbine, multiple-blade drills by headpiece for removing the decayed dentine and, after cleaning and control of bleeding with cotton pellets with saline solution,RM-GIC (3M ESPE, USA) light-hardening paste was placed gently on the exposed part of the pulp and cavity floor next final restoration with composite z350 flow able and p60 (3M ESPE, USA).
- Diode 808 nm laser-assisted group: 2. Group B : Five teeth cavities were prepared as the same with group one with traditional rotating instruments, hemostatic and cavities sterilization were achieved by a diode 808 nm (Picasso- AMD, USA) laser using following parameters:
  * Hemostatic: 1.5 W, CW, fiber diameter 400µm, in contact, 2s per 1mm, vertical and horizontal scanning movement on exposure site.
  * Cavity sterilization: 1W, CW, fiber diameter 400µm, in contact, 2mm per s, circular movement.
  After hemostatic and cavity sterilization, RM-GIC (3M ESPE, USA) light-hardening paste was placed on the exposed part of the pulp and cavity floor next final restoration with composite z350 flow able and p60 (3M ESPE, USA).

SUMMARY:
The purpose of this study was to compare the conventional and diode 808 nm laser-assisted techniques in direct pulp capping in permanent teeth .The present study was based on a series of ten clinical studies with pulp exposure caused by carious lesions.The hypothesis of this paper was laser supported direct pulp cap-ping has proven effectiveness by its capacity to stimulate reparative dentine formation by pulp cells, de-contamination ability of irradiated areas, its ability in the fast and better haemostatic, and pain reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent teeth with deep caries
2. Vitality of teeth
3. No peri-apical radiographic changes
4. Acceptance research program

Exclusion Criteria:

1. Symptoms
2. Peri-apical radiographic changes
3. No stopped bleeding within 3 minutes after exposure
4. No acceptance study program

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study was carried out on 10 patients, aged between 12 and 40 years, with an average age of 26 years, who underwent conservative treatment for deep caries of permanent teeth (2 anterior and 8 posterior).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Maintenance of teeth vitality was be measured via thermal tests also by radiographic. | up to 12 months
  Given low success rate of conventional methods, new techniques as laser-assisted need to be developed.The outcome measure of this study was maintenance of teeth vitality with carious exposed via tertiary dentine formation.the tertiary dentine formation during the time of study was assessed radiological. Therefore vitality of the teeth was depend on dentine formation that was measured periodically in 1,6 and 12 months.